CLINICAL TRIAL: NCT05107141
Title: Ridge Preservation in Molar Sites Comparing Xenograft Versus Mineralized Freeze-dried Bone Allograft: a Randomized Clinical Trial
Brief Title: Ridge Preservation in Molar Sites Comparing Xenograft Versus Mineralized Freeze-dried Bone Allograft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Collaborators: BioHorizons, Inc. (Industry); Geistlich Pharma AG (Industry); Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Principal Investigator, Desire Abellán Iñiguez, Principal investigator, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013-M-PER-ECL-2013-04
Record Dates: First submitted 2021-10-10; First posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Alveolar Ridge Preservation
Keywords: alveolar ridge preservation; molars; xenograft; allograft
MeSH Terms: interventions — Bone Transplantation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- xenograft and a collagen membrane (Active Comparator)
  Interventions: Procedure: Ridge preservation; Device: bone graft plus a collagen membrane
- allograft and a collagen membrane (Active Comparator)
  Interventions: Procedure: Ridge preservation; Device: bone graft plus a collagen membrane

INTERVENTIONS:
Procedure: Ridge preservation — Ridge preservation in molar areas using a xenograft or an allograft in combination with a barrier collagen membrane
Device: bone graft plus a collagen membrane

SUMMARY:
The objectives of the present investigation are; to compare the dimensional changes and the histological composition after the use of an allograft or xenograft and a resorbable membrane in ridge preservation in molar sites, to evaluate the influence of bone plates thickness on dimensional changes and the effectiveness of ridge preservation in limiting the need of sinus elevation.

DETAILED DESCRIPTION:
Twenty-four patients in need of maxillary or mandibular molar extraction and subsequent implant placement were included and randomly assigned to a group; allograft or xenograft, plus a collagen membrane. Cone Beam Computed Tomographies were obtained after molar extraction and after five months. A bone sample was harvested at the time of implant placement and analysed by histomorphometry.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, over 18 years old.
* In need of removal of a maxillary or mandibular molar first or second molar.
* The molars to be extracted had to be bordered by at least one tooth.
* The molars had to have a presence of > 2 mm of keratinized gingiva and three intact bony walls.
* A dehiscence on the fourth wall, if any, had to be equal or less than 2 mm in height.
* Only one extraction per patient was accepted.

Exclusion Criteria:

* Acute periodontal or periapical infection.
* Pregnancy or lactancy.
* Smokers of more than 10 cigarettes per day.
* Previous adverse reactions to the biomaterials used in the study.
* Metabolic diseases affecting the mechanism of bone remodelling.
* Medications or treatments taken in the last twelve months and known to affect bone "turnover".
* Patients with poor plaque control -more than 20% (O'Leary, Drake, Naylor, 1972).
* Patients with absence of periodontal health maintenance or postoperative recommendations compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-12-09 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2019-06-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of ridge dimensional changes following ridge preservation in molar sites comparing the use of freeze dried bone allograft (FDBA) or xenograft (DBBM), and a resorbable membrane. | 5 months
  To evaluate dimensional changes, the initial (CBCT1) and 5 months (CBCT2) CBCT images were processed and superimposed with the use of a specialized software image Simplant® O&O (Denstply Sirona, Charlotte, NC, USA).
  Measurements were expressed in millimeters (mm) and percentages showing changes in ridge width at 1mm, 3mm and 5mm from the bone crest.
  The height of the buccal, and lingual bone crest was assessed, as well as the heigh in the central are of the socket.

SECONDARY OUTCOMES:
Evaluate the influence of buccal or lingual bone thickness on bone ridge changes | 5 months
  The width of the buccal and lingual bone plates was evaluated, by CBCT analysis, at 1mm, 3mm and 5mm to evaluate any correlation with bone dimensional changes after 5 months.
  Data was expressed in milimeters.
Evaluate the histologic composition of the regenerated areas after the use of freeze dried bone allograft (FDBA) or xenograft (DBBM), and a resorbable membrane. | 5 months
  The histomorphometric analysis was performed by the use of a specific software image (Image J®, Image Processing and Analysis in Java) and the areas occupied by vital bone (VB), non-mineralized connective tissue (NMCT) and graft particles (GP) were evaluated. The analysis of each tissue volume was expressed in percentages (%)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Nart Molina, Study Director — Universitat Internacional de Catalunya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Avila-Ortiz G, Chambrone L, Vignoletti F. Effect of alveolar ridge preservation interventions following tooth extraction: A systematic review and meta-analysis. J Clin Periodontol. 2019 Jun;46 Suppl 21:195-223. doi: 10.1111/jcpe.13057. Erratum In: J Clin Periodontol. 2020 Jan;47(1):129. doi: 10.1111/jcpe.13212. PMID 30623987
- [Background] Nart J, Barallat L, Jimenez D, Mestres J, Gomez A, Carrasco MA, Violant D, Ruiz-Magaz V. Radiographic and histological evaluation of deproteinized bovine bone mineral vs. deproteinized bovine bone mineral with 10% collagen in ridge preservation. A randomized controlled clinical trial. Clin Oral Implants Res. 2017 Jul;28(7):840-848. doi: 10.1111/clr.12889. Epub 2016 Jun 22. PMID 27335267
- [Background] Tonetti MS, Jung RE, Avila-Ortiz G, Blanco J, Cosyn J, Fickl S, Figuero E, Goldstein M, Graziani F, Madianos P, Molina A, Nart J, Salvi GE, Sanz-Martin I, Thoma D, Van Assche N, Vignoletti F. Management of the extraction socket and timing of implant placement: Consensus report and clinical recommendations of group 3 of the XV European Workshop in Periodontology. J Clin Periodontol. 2019 Jun;46 Suppl 21:183-194. doi: 10.1111/jcpe.13131. PMID 31215112
- [Background] Walker CJ, Prihoda TJ, Mealey BL, Lasho DJ, Noujeim M, Huynh-Ba G. Evaluation of Healing at Molar Extraction Sites With and Without Ridge Preservation: A Randomized Controlled Clinical Trial. J Periodontol. 2017 Mar;88(3):241-249. doi: 10.1902/jop.2016.160445. Epub 2016 Oct 27. PMID 27788625
- [Background] Duong M, Mealey BL, Walker C, Al-Harthi S, Prihoda TJ, Huynh-Ba G. Evaluation of healing at molar extraction sites with and without ridge preservation: A three-arm histologic analysis. J Periodontol. 2020 Jan;91(1):74-82. doi: 10.1002/JPER.19-0237. Epub 2019 Aug 11. PMID 31355447